CLINICAL TRIAL: NCT04469842
Title: A Prospective, Randomized, Controlled Pilot Study of Early-Use Long Acting Tacrolimus (Envarsus XR) in Lung Transplant Recipients
Brief Title: Early Use of Long-acting Tacrolimus in Lung Transplant Recipients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Anil Trindade, Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VEL-IIS-2020-085
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Lung Transplant; Complications
Keywords: Lung Transplantation; Calcineurin inhibitor; LCP-tacrolimus (Envarsus XR); Calcineurin-inhibitor nephrotoxicity (CIN)
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Prednisone; Azathioprine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunosuppression with Extended-Release Tacrolimus (Experimental): LCP-tacrolimus administered daily to target a goal trough level of 10-14 ng/mL x 7 months (with Mycophenolate mofetil and prednisone).
  Additional standard immunosuppression with either mycophenolate mofetil (500-1500mg twice daily) OR Azathioprine (up to 2mg/kg daily) AND Prednisone (5-10mg daily) will be administered.
  Interventions: Drug: Tacrolimus Extended Release Oral Tablet [Envarsus]; Drug: Mycophenolate Mofetil Hydrochloride; Drug: Prednisone; Drug: Azathioprine
- Immunosuppression with Intermediate Release Tacrolimus (Active Comparator): IR-tacrolimus administered twice daily to target a goal trough level of 10-14 ng/mL x 7 months (with Mycophenolate mofetil and prednisone). This is currently the standard of care at Vanderbilt University Medical Center and most other lung transplant centers (ISHLT Registry 2019).
  Additional standard immunosuppression with either mycophenolate mofetil (500-1500mg twice daily) OR Azathioprine (up to 2mg/kg daily) AND Prednisone (5-10mg daily) will be administered.
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate Mofetil Hydrochloride; Drug: Prednisone; Drug: Azathioprine

INTERVENTIONS:
Drug: Tacrolimus Extended Release Oral Tablet [Envarsus] — Immunosuppression regimen with Tacrolimus Extended Release as the backbone.
  Other Names: Envarsus XR
  Arms: Immunosuppression with Extended-Release Tacrolimus
Drug: Tacrolimus — Standard Immunosuppression regimen with Intermediate-Release Tacrolimus.
  Other Names: Intermediate Release Tacrolimus; Prograf; FK506
  Arms: Immunosuppression with Intermediate Release Tacrolimus
Drug: Mycophenolate Mofetil Hydrochloride — Standard immunosuppression of the anti-proliferative class.
  Other Names: MMF; CellCept
Drug: Prednisone — Standard immunosuppression (corticosteroid class).
  Other Names: Deltasone
Drug: Azathioprine — Standard immunosuppression of the anti-proliferative class.
  Other Names: Imuran

SUMMARY:
Lung transplantation is a life-saving therapy for patients with advanced lung disease, however, necessitates the use of life-long immunosuppressive therapy for the prevention of acute and chronic rejection. The backbone of immunosuppression is the calcineurin-inhibitor class, with tacrolimus being the preferred drug due to its potency and improved side-effect profile. Nevertheless, tacrolimus is associated with several side effects including increased risk for infection and malignancy, tremors, headaches, seizures, hypertension, leukopenia and renal dysfunction. In fact, by 6 months post-transplant, 50% of patients will have a 50% decline in eGFR and by 5 years post-transplant ~10% of patients will have advanced renal disease that may require renal replacement therapy and/or kidney transplantation. Tacrolimus induces a nephropathy in two ways- acute calcineurin inhibitor nephrotoxicity (CIN) is mediated by afferent arteriolar vasoconstriction, whereas chronic CIN is due to interstitial nephritis and fibrosis. Immunosuppressive regimens that spare or dose-reduce calcineurin inhibitors have been shown to have a modest impact on preserving renal function, but are limited by timing. Although most studies support implementing renal preserving protocols early on, this is balanced by the potential for acute cellular rejection, antibody mediated rejection and anastomotic dehiscence.

Long-acting Tacrolimus (LCP-tacrolimus) may have the potential to bridge the balance of providing potent immunosuppression, while sparing renal function, due to the better systemic dose levels and improved concentration/dose ration achieved with it compared to IR-tacrolimus, evidenced in the renal transplant population. There is limited experience with LCP-tacrolimus in lung transplantation. Several case reports chronicling the late conversion from IR-tacrolimus to LCP-tacrolimus due to absorption issues or side-effect intolerance, have demonstrated safety and tolerability. The investigators seek to determine whether early use of LCP-tacrolimus in lung transplant recipients following the index hospitalization is acceptable, and propose a single-center prospective, randomized, controlled pilot study of early-use LCP-tacrolimus in lung transplant recipients to assess safety, tolerability and side-effects of LCP-tacrolimus.

DETAILED DESCRIPTION:
Lung transplantation is a life-saving therapy for patients with end-stage lung disease refractory to medical treatment, providing an improvement in both survival and quality of life.[1,2] Despite the benefits, patients are at risk for myriad side effects including infection, malignancy, neurologic complications (headache, tremor, seizures), gastrointestinal distress and renal failure, to name a few.[3] Many of these are related to the requisite need for life-long immunosuppression. Current standard immunosuppressive regimens for lung transplant recipients include calcineurin inhibitors (tacrolimus preferred over cyclosporine), antiproliferative agents (mycophenolate mofetil vs. azathioprine) and corticosteroids; calcineurin inhibitors serve as the backbone of immunosuppression.[4] Renal dysfunction is perhaps the most prevalent complication after lung transplantation, affecting up to 90% of post-transplant recipients.[5] By 5-year post-transplant, ~8% of patients may require renal replacement therapy and/or renal transplantation.[6] Renal dysfunction tends to occur early on in the post-transplant period. Monnier and colleagues showed in a single-center analysis that the incidence of acute kidney injury within the index hospitalization was ~75%; the median loss of glomerular function within the first year was ~45%.[7] Moreover, Canales and colleagues showed that >55% of patients in a cohort of 219 lung transplant recipients had a doubling of their pre-transplant serum creatinine, the majority occurring within the first year post-transplant.[8] Early renal dysfunction in lung transplant recipients is associated with a poor overall prognosis. Broelkroleof and colleagues demonstrated that loss of renal function within he first month post-transplant is predictive of chronic kidney disease.[9] Moreover, chronic kidney disease is associated with a five times increased risk of mortality.[5] Perhaps the greatest contributor to the development of CKD in solid-organ transplant recipients are the calcineurin inhibitors (CNIs).[10] CNIs cause renal compromise (calcineurin inhibitor nephropathy, CIN) via acute and chronic mechanisms. Acute CIN is due to potent vasoconstriction of afferent arterioles in the kidney, resulting in ischemia.[11,12] Chronic CIN is thought to be largely mediated by interstitial fibrosis as the end-result of arteriolar sclerosis, oxygen free-radical injury, and upregulation of pro-fibrotic pathways including PDGF, renin-angiotensin-aldosterone signaling, TGFB and matrix metalloproteinase-9.[11,13] Attempts at utilizing CNI-free or CNI-reduced regimens in the lung transplantation population has been understudied and/or unsuccessful to date. Belatacept, a CTLA4-fusion molecule that prevents CD28-mediated co-stimulation to activate T-lymphocytes, has been well-studied in renal transplantation as an alternative to CNIs. The BENEFIT Trial, a phase III clinical study of Belatacept vs. Cyclosporine in renal transplant recipients, demonstrated improvement in patient and allograft survival, and mean eGFR (~70 cc/min vs ~45cc/min) at seven years. However, rates of biopsy proven acute cellular rejection were twice as much with Belatacept.[14] Case reports of Belatacept as rescue therapy in lung transplant recipients intolerant of CNIs are mixed; there are reports of increased ACR and fulminant acute respiratory distress syndrome.[15,16] The mTOR inhibitor class of immunosuppression has also been incorporated into regimens in an effort to ameliorate CNI-toxicity. Villanueva and colleagues assessed outcomes of conversion to Sirolimus and reduced Tacrolimus in 49 patients with bronchiolitis obliterans syndrome (chronic rejection) or CNI-intolerance; there was no difference in renal function one year following sirolimus initiation.[17] Conversely, Shitrit and colleagues demonstrated that sirolimus plus low-dose tacrolimus led to an improvement in GFR of 10 mL/min, compared to control maintenance immunosuppression in a pilot study of sixteen lung allograft recipients.[18] More recently, Gottlieb and colleagues demonstrated that conversion to quadruple immunosuppression therapy with low-dose CNI (target tacrolimus trough 3-5) led to improvements in eGFR of 10cc/mL compared to standard immunosuppression (tacrolimus trough >5). There was no considerable difference in biopsy-proven acute rejection, chronic rejection and death.[20] The conversion for those in the 4-drug experimental group occurred on average 11 months following transplant, which may account for the muted benefit; perhaps an earlier change in immunosuppression management would have led to more clinically significant results. Notably, discontinuation rates of sirolimus in case reports are variable, with most studies reporting a 20-80% discontinuation rate due to gastrointestinal distress, pneumonitis, thrombocytopenia, etc., making the mTOR inhibitor class less appealing.[19] It is apparent that changes to immunosuppression management earlier in the post-transplant period are ideal to see a maximum benefit in preserved renal function.9 However, this is complicated by the concerns for acute cellular rejection, which has a peak incidence at 6 months post-lung transplantation.[21,22] Acute cellular rejection is a leading risk factor for the development of chronic lung allograft dysfunction (CLAD, chronic rejection).[23] Hence any dose reduction in CNI or the use of an agent associated with ACR (Belatacept) is less desirable within the first few months post-transplant.

Given the preference to utilize a CNI-based regimen early-post transplant but still minimize nephrotoxic effects, the investigators seek to determine whether the early use of long acting tacrolimus, LCP-Tacrolimus (LCP-tacro, Envarsus XR, Veloxis Pharmaceuticals), results in improved renal function compared to intermediate release tacrolimus (IR-tacrolimus, IR-tacro). Anecdotally, LCP-tacro has been used in lung transplant recipients as an alternative agent for those with debilitating headache or tremor. Early use of LCP-tacro has not been widely adopted due to perceptions associated with ability to closely titrate trough levels and cost. However, early use of LCP-tacro may provide several benefits. As a long-acting formulation, LCP-tacro allows for daily dosing. Moreover, LCP-tacro has greater absorption and bioavailability, leading to decreased swings in peak and trough concentrations; frequent fluctuations in serum tacrolimus levels potentiates afferent arteriolar vasoconstriction.[24] A steady state of systemic tacrolimus trough levels is desirable, since tacrolimus metabolism is directly related to nephrotoxicity.[25] The use of LCP-Tacro has been studied in renal transplant recipients. Langone and colleagues identified that LCP-tacrolimus compared to IR-tacrolimus was associated with improved tremor incidence and quality of life.[1] Rostaing and colleagues demonstrated that the use of LCP-tacro compared to intermediate tacrolimus was non-inferior in terms of combined death, allograft failure, biopsy-proven acute rejection and loss to follow-up. However, the use of LCP-tacro was associated with a significant reduction in total daily dose, and a 30% reduction in peak dose, without an increase in biopsy proven acute rejection episodes. Although not a prospective end-point, there was no significant impact on renal function.[26] In other studies, though, higher concentration/ drug (C/D) ratios for tacrolimus are associated with an improved renal safety profile.[27] It is conceivable that a clinical benefit of LCP-tacro over IR-tacro may be better manifested in clinical arenas that require higher target tacrolimus trough levels, such as lung allograft recipients, where initial post-transplant targets can be as high as 12-15 ng/mL, compared to renal transplantation where target trough levels are a relatively conservative 4-8 ng/mL.[2, 3] The experience of LCP-tacrolimus in the realm of lung transplantation is limited. Murakoezy and colleagues studied 53 patients that were converted from short-acting Tacrolimus to long-acting Envarsus. Conversion was performed at an average 3.6 years post-transplant. Ten patients were switched back due to side-effects (unknown), though the remainder tolerated conversion without complication. Ahmed and colleagues demonstrated feasibility in using long-acting Tacrolimus in 8 patients that were unable to achieve sufficient therapeutic levels with a short-acting formulation due to suspected polymorphisms of CYP3A4/3A5.[28] McCurry and colleagues assessed safety and feasibility of LCP-tacrolimus in a retrospective analysis of 18 lung transplant recipients. They found that patients on LCP-tacro had a 27% reduction in total dose. No patients experienced any adverse effects. Moreover, 2/18 patients had an improvement in tremors and headache.[29] Given the limited experience with of LCP-tacrolimus in lung transplant populations, the investigators propose a prospective, randomized, controlled pilot study to assess the safety, tolerability, and side-effect profile of early use LCP-tacro within the first 9 months post-transplantation. It is hypothesized that the early use of LCP-tacro in lung transplant recipients is safe and tolerable, and associated with an improved side-effect profile compared to patients treated with standard IR-tacro.

ELIGIBILITY:
Inclusion Criteria:

* Status-post single or bilateral lung transplantation
* Participant is able to give informed consent for participation in the study.
* Male or female age 18 years or above.
* Actively receives care at VUMC and is adherent with medical therapies.

Exclusion Criteria:

* History of prior organ transplantation
* History of tacrolimus use prior to transplantation
* Intolerance of tacrolimus (that precludes use)
* Having DSA pre-transplant (Positive virtual crossmatch)
* Active infection with Hepatitis B or C
* Active infection with Human Immunodeficiency Virus (HIV)
* Baseline AST / ALT > three times upper limit normal
* Primary graft dysfunction grade 3 at 72 hours
* Acute kidney injury during index hospitalization that does not resolve to two times the pre-transplant baseline value.
* Contraindication to PO (per os) intake of medications
* Impaired GI absorption (defined as sublingual administration of IR-tacro)
* History of frequent headaches
* Seizure history
* Cannot provide consent (at least verbally)
* Pregnancy or breast-feeding
* Participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 6 months
  Composite of mortality, allograft failure, potential drug induced liver injury, supra-therapeutic trough levels (>20 ng/mL), sub-therapeutic trough levels (<5 ng/mL), seizures, encephalopathy, thrombotic microangiopathy and serious hyperkalemia associated with use of LCP-tacrolimus, compared to matched historical controls administered IR-tacrolimus.

SECONDARY OUTCOMES:
Median change in eGFR at 9 months post-transplant. | 9 months
  Median change in eGFR from study start to 9 months post-transplantation with patients administered LCP-tacrolimus compared to IR-tacrolimus.
Headache frequency and severity | 9 months
  Quality of life related to headache frequency and severity using the Headache Impact Tool (HIT-6).
Quality of life related to tremor | 9 months
  Quality of life related to tremor as measured by the QUEST tool.
Incidence of acute cellular rejection | 9 months
  Incidence of acute cellular rejection (>= A1) or lymphocytic bronchiolitis (>= B1R)
Incidence of de novo donor-specific anti-HLA antibodies | 9 months
  Incidence of de novo donor-specific anti-HLA antibodies (MFI > 1500) within the first 9 months post-transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Anil J Trindade, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rana A, Gruessner A, Agopian VG, Khalpey Z, Riaz IB, Kaplan B, Halazun KJ, Busuttil RW, Gruessner RW. Survival benefit of solid-organ transplant in the United States. JAMA Surg. 2015 Mar 1;150(3):252-9. doi: 10.1001/jamasurg.2014.2038. PMID 25629390
- [Background] Singer JP, Katz PP, Soong A, Shrestha P, Huang D, Ho J, Mindo M, Greenland JR, Hays SR, Golden J, Kukreja J, Kleinhenz ME, Shah RJ, Blanc PD. Effect of Lung Transplantation on Health-Related Quality of Life in the Era of the Lung Allocation Score: A U.S. Prospective Cohort Study. Am J Transplant. 2017 May;17(5):1334-1345. doi: 10.1111/ajt.14081. Epub 2017 Jan 3. PMID 27743488
- [Background] Lyu DM, Zamora MR. Medical complications of lung transplantation. Proc Am Thorac Soc. 2009 Jan 15;6(1):101-7. doi: 10.1513/pats.200808-077GO. PMID 19131535
- [Background] Scheffert JL, Raza K. Immunosuppression in lung transplantation. J Thorac Dis. 2014 Aug;6(8):1039-53. doi: 10.3978/j.issn.2072-1439.2014.04.23. PMID 25132971
- [Background] Ojo AO, Held PJ, Port FK, Wolfe RA, Leichtman AB, Young EW, Arndorfer J, Christensen L, Merion RM. Chronic renal failure after transplantation of a nonrenal organ. N Engl J Med. 2003 Sep 4;349(10):931-40. doi: 10.1056/NEJMoa021744. PMID 12954741
- [Background] Chambers DC, Cherikh WS, Harhay MO, Hayes D Jr, Hsich E, Khush KK, Meiser B, Potena L, Rossano JW, Toll AE, Singh TP, Sadavarte A, Zuckermann A, Stehlik J; International Society for Heart and Lung Transplantation. The International Thoracic Organ Transplant Registry of the International Society for Heart and Lung Transplantation: Thirty-sixth adult lung and heart-lung transplantation Report-2019; Focus theme: Donor and recipient size match. J Heart Lung Transplant. 2019 Oct;38(10):1042-1055. doi: 10.1016/j.healun.2019.08.001. Epub 2019 Aug 8. No abstract available. PMID 31548030
- [Background] Canales M, Youssef P, Spong R, Ishani A, Savik K, Hertz M, Ibrahim HN. Predictors of chronic kidney disease in long-term survivors of lung and heart-lung transplantation. Am J Transplant. 2006 Sep;6(9):2157-63. doi: 10.1111/j.1600-6143.2006.01458.x. Epub 2006 Jul 6. PMID 16827787
- [Background] Broekroelofs J, Navis GJ, Stegeman CA, van der Bij W, de Boer WJ, de Zeeuw D, de Jong PE. Long-term renal outcome after lung transplantation is predicted by the 1-month postoperative renal function loss. Transplantation. 2000 Apr 27;69(8):1624-8. doi: 10.1097/00007890-200004270-00017. PMID 10836372
- [Background] Bloom RD, Reese PP. Chronic kidney disease after nonrenal solid-organ transplantation. J Am Soc Nephrol. 2007 Dec;18(12):3031-41. doi: 10.1681/ASN.2007040394. PMID 18039925
- [Background] Naesens M, Kuypers DR, Sarwal M. Calcineurin inhibitor nephrotoxicity. Clin J Am Soc Nephrol. 2009 Feb;4(2):481-508. doi: 10.2215/CJN.04800908. PMID 19218475
- [Background] Hoorn EJ, Walsh SB, McCormick JA, Zietse R, Unwin RJ, Ellison DH. Pathogenesis of calcineurin inhibitor-induced hypertension. J Nephrol. 2012 May-Jun;25(3):269-75. doi: 10.5301/jn.5000174. PMID 22573529
- [Background] Gaston RS. Chronic calcineurin inhibitor nephrotoxicity: reflections on an evolving paradigm. Clin J Am Soc Nephrol. 2009 Dec;4(12):2029-34. doi: 10.2215/CJN.03820609. Epub 2009 Oct 22. PMID 19850771
- [Background] Vincenti F, Rostaing L, Grinyo J, Rice K, Steinberg S, Gaite L, Moal MC, Mondragon-Ramirez GA, Kothari J, Polinsky MS, Meier-Kriesche HU, Munier S, Larsen CP. Belatacept and Long-Term Outcomes in Kidney Transplantation. N Engl J Med. 2016 Jan 28;374(4):333-43. doi: 10.1056/NEJMoa1506027. PMID 26816011
- [Background] Timofte I, Terrin M, Barr E, Sanchez P, Kim J, Reed R, Britt E, Ravichandran B, Rajagopal K, Griffith B, Pham S, Pierson RN 3rd, Iacono A. Belatacept for renal rescue in lung transplant patients. Transpl Int. 2016 Apr;29(4):453-63. doi: 10.1111/tri.12731. Epub 2016 Feb 8. PMID 26678245
- [Background] Iasella CJ, Winstead RJ, Moore CA, Johnson BA, Feinberg AT, Morrell MR, Hayanga JWA, Lendermon EA, Zeevi A, McDyer JF, Ensor CR. Maintenance Belatacept-Based Immunosuppression in Lung Transplantation Recipients Who Failed Calcineurin Inhibitors. Transplantation. 2018 Jan;102(1):171-177. doi: 10.1097/TP.0000000000001873. PMID 28691954
- [Background] Villanueva J, Boukhamseen A, Bhorade SM. Successful use in lung transplantation of an immunosuppressive regimen aimed at reducing target blood levels of sirolimus and tacrolimus. J Heart Lung Transplant. 2005 Apr;24(4):421-5. doi: 10.1016/j.healun.2004.01.014. PMID 15797743
- [Background] Shitrit D, Rahamimov R, Gidon S, Bakal I, Bargil-Shitrit A, Milton S, Kramer MR. Use of sirolimus and low-dose calcineurin inhibitor in lung transplant recipients with renal impairment: results of a controlled pilot study. Kidney Int. 2005 Apr;67(4):1471-5. doi: 10.1111/j.1523-1755.2005.00224.x. PMID 15780099
- [Background] Gottlieb J, Neurohr C, Muller-Quernheim J, Wirtz H, Sill B, Wilkens H, Bessa V, Knosalla C, Porstner M, Capusan C, Struber M. A randomized trial of everolimus-based quadruple therapy vs standard triple therapy early after lung transplantation. Am J Transplant. 2019 Jun;19(6):1759-1769. doi: 10.1111/ajt.15251. Epub 2019 Feb 5. PMID 30615259
- [Background] Martinu T, Chen DF, Palmer SM. Acute rejection and humoral sensitization in lung transplant recipients. Proc Am Thorac Soc. 2009 Jan 15;6(1):54-65. doi: 10.1513/pats.200808-080GO. PMID 19131531
- [Background] Martinu T, Pavlisko EN, Chen DF, Palmer SM. Acute allograft rejection: cellular and humoral processes. Clin Chest Med. 2011 Jun;32(2):295-310. doi: 10.1016/j.ccm.2011.02.008. Epub 2011 Mar 25. PMID 21511091
- [Background] Husain AN, Siddiqui MT, Holmes EW, Chandrasekhar AJ, McCabe M, Radvany R, Garrity ER. Analysis of risk factors for the development of bronchiolitis obliterans syndrome. Am J Respir Crit Care Med. 1999 Mar;159(3):829-33. doi: 10.1164/ajrccm.159.3.9607099. PMID 10051258
- [Background] Gaber AO, Alloway RR, Bodziak K, Kaplan B, Bunnapradist S. Conversion from twice-daily tacrolimus capsules to once-daily extended-release tacrolimus (LCPT): a phase 2 trial of stable renal transplant recipients. Transplantation. 2013 Jul 27;96(2):191-7. doi: 10.1097/TP.0b013e3182962cc1. PMID 23715050
- [Background] Tholking G, Fortmann C, Koch R, Gerth HU, Pabst D, Pavenstadt H, Kabar I, Husing A, Wolters H, Reuter S, Suwelack B. The tacrolimus metabolism rate influences renal function after kidney transplantation. PLoS One. 2014 Oct 23;9(10):e111128. doi: 10.1371/journal.pone.0111128. eCollection 2014. PMID 25340655
- [Background] Rostaing L, Bunnapradist S, Grinyo JM, Ciechanowski K, Denny JE, Silva HT Jr, Budde K; Envarsus Study Group. Novel Once-Daily Extended-Release Tacrolimus Versus Twice-Daily Tacrolimus in De Novo Kidney Transplant Recipients: Two-Year Results of Phase 3, Double-Blind, Randomized Trial. Am J Kidney Dis. 2016 Apr;67(4):648-59. doi: 10.1053/j.ajkd.2015.10.024. Epub 2015 Dec 22. PMID 26717860
- [Background] Langone A, Steinberg SM, Gedaly R, Chan LK, Shah T, Sethi KD, Nigro V, Morgan JC; STRATO Investigators. Switching STudy of Kidney TRansplant PAtients with Tremor to LCP-TacrO (STRATO): an open-label, multicenter, prospective phase 3b study. Clin Transplant. 2015 Sep;29(9):796-805. doi: 10.1111/ctr.12581. Epub 2015 Aug 6. PMID 26113208
- [Background] Baker RJ, Mark PB, Patel RK, Stevens KK, Palmer N. Renal association clinical practice guideline in post-operative care in the kidney transplant recipient. BMC Nephrol. 2017 Jun 2;18(1):174. doi: 10.1186/s12882-017-0553-2. PMID 28571571
- [Background] Troster AI, Pahwa R, Fields JA, Tanner CM, Lyons KE. Quality of life in Essential Tremor Questionnaire (QUEST): development and initial validation. Parkinsonism Relat Disord. 2005 Sep;11(6):367-73. doi: 10.1016/j.parkreldis.2005.05.009. PMID 16103000
- [Background] Yang M, Rendas-Baum R, Varon SF, Kosinski M. Validation of the Headache Impact Test (HIT-6) across episodic and chronic migraine. Cephalalgia. 2011 Feb;31(3):357-67. doi: 10.1177/0333102410379890. Epub 2010 Sep 6. PMID 20819842
- [Background] Sikma MA, van Maarseveen EM, Donker DW, Meulenbelt J. Letter to the editor: "Immunosuppressive drug therapy--biopharmaceutical challenges and remedies". Expert Opin Drug Deliv. 2015;12(12):1955-6; discussion 1956-7. doi: 10.1517/17425247.2015.1106687. Epub 2015 Nov 7. No abstract available. PMID 26549727
- [Background] Bunnapradist S, Ciechanowski K, West-Thielke P, Mulgaonkar S, Rostaing L, Vasudev B, Budde K; MELT investigators. Conversion from twice-daily tacrolimus to once-daily extended release tacrolimus (LCPT): the phase III randomized MELT trial. Am J Transplant. 2013 Mar;13(3):760-9. doi: 10.1111/ajt.12035. Epub 2012 Dec 21. PMID 23279614
- [Background] Kotloff RM, Ahya VN. Medical complications of lung transplantation. Eur Respir J. 2004 Feb;23(2):334-42. doi: 10.1183/09031936.03.00043403. PMID 14979513
- [Background] Ferrari U, Empl M, Kim KS, Sostak P, Forderreuther S, Straube A. Calcineurin inhibitor-induced headache: clinical characteristics and possible mechanisms. Headache. 2005 Mar;45(3):211-4. doi: 10.1111/j.1526-4610.2005.05046.x. PMID 15836594
- [Background] Maggioni F, Mantovan MC, Rigotti P, Cadrobbi R, Mainardi F, Mampreso E, Ermani M, Cortelazzo S, Zanchin G. Headache in kidney transplantation. J Headache Pain. 2009 Dec;10(6):455-60. doi: 10.1007/s10194-009-0148-9. Epub 2009 Aug 27. PMID 19711000
- [Background] Waikar SS, Rebholz CM, Zheng Z, Hurwitz S, Hsu CY, Feldman HI, Xie D, Liu KD, Mifflin TE, Eckfeldt JH, Kimmel PL, Vasan RS, Bonventre JV, Inker LA, Coresh J; Chronic Kidney Disease Biomarkers Consortium Investigators. Biological Variability of Estimated GFR and Albuminuria in CKD. Am J Kidney Dis. 2018 Oct;72(4):538-546. doi: 10.1053/j.ajkd.2018.04.023. Epub 2018 Jul 18. PMID 30031564
- [Background] Levine DJ, Glanville AR, Aboyoun C, Belperio J, Benden C, Berry GJ, Hachem R, Hayes D Jr, Neil D, Reinsmoen NL, Snyder LD, Sweet S, Tyan D, Verleden G, Westall G, Yusen RD, Zamora M, Zeevi A. Antibody-mediated rejection of the lung: A consensus report of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2016 Apr;35(4):397-406. doi: 10.1016/j.healun.2016.01.1223. Epub 2016 Feb 10. PMID 27044531
- [Background] Ahmed SK, Seethamraju H. CYP3A5 Polymorphisms and Conversion to Once-Daily, Extended-Release Tacrolimus in Lung Transplant (LTx). J Heart Lung Transplant. 2020; 39(4): S505.
- [Result] Monnier A, Kummel T, Collage O, et al. Prevalence of Acute and Chronic Renal Failure After Lung Transplantation. In. Vol 34. Journal Heart Lung Transplantation 2015:S261.
- [Result] McCurry KA,Fitzgerald LJ, Chan JM, Jia S. Conversion from Tacrolimus IR (Twice Daily) or Cyclosporine to Tacrolimus XR (Envarsus®, Once Daily) in Lung Transplant Recipients. J Heart Lung Transplant. 2020; 39(4): S505